CLINICAL TRIAL: NCT00022412
Title: Phase II Open Label, Multi-Center Clinical Trial Of Modulation Of Intermediate Endpoint Biomarkers By 1x-Hydroxyvitamin D2 In Patients With Clinically Localized Prostate Cancer And High Grade PIN
Brief Title: Doxercalciferol Before Surgery in Treating Localized Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO99802; P30CA014520 (NIH); WCCC-CO-99802; NCI-N01-CN-95130; WCCC-CO-2000169; NCI-P01-0188; CDR0000068813 (Other); 2000-595 (Other: Institutional Review Board)
Record Dates: First submitted 2001-08-10; First posted 2003-01-27 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2016-10

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage II prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 1 alpha-hydroxyergocalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Observation, then prostatectomy (Placebo Comparator): Arm 2: Patients undergo observation for 28 days. Patients then undergo prostatectomy.
  Interventions: Procedure: conventional surgery
- Doxercalciferol once daily for 28 days (Active Comparator): Dietary supplement once daily to treat prostate cancer for 28 days
  Interventions: Dietary Supplement: doxercalciferol

INTERVENTIONS:
Dietary Supplement: doxercalciferol — Arm 1: Patients receive doxercalciferol once daily for 28 days. Patients then undergo prostatectomy.
  Other Names: Localized adenocarcinoma of the prostate
  Arms: Doxercalciferol once daily for 28 days
Procedure: conventional surgery — Procedure: Prostatectomy for prostate cancer
  Other Names: Prostatectomy - no dietary supplement
  Arms: Observation, then prostatectomy

SUMMARY:
RATIONALE: Doxercalciferol may be an effective way to treat localized prostate cancer before surgery.

PURPOSE: Randomized phase II trial to study the effectiveness of giving doxercalciferol before surgery in treating patients who have localized prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether doxercalciferol modulates intermediate endpoint biomarkers in the development of prostate cancer in patients with localized prostate cancer.
* Assess the toxicity of this drug in these patients.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are randomized to one of 2 arms.

* Arm I: Patients receive doxercalciferol once daily for 28 days. Patients then undergo prostatectomy.
* Arm II: Patients undergo observation for 28 days. Patients then undergo prostatectomy.

PROJECTED ACCRUAL: A total of 60 patients (30 per arm) will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed localized adenocarcinoma of the prostate
* Candidate for prostatectomy

PATIENT CHARACTERISTICS:

Age:

* 21 and over

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 4,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.4 mg/dL
* AST no greater than 3 times normal

Renal:

* Creatinine no greater than 2.0 mg/dL
* Calcium no greater than 10.2 mg/dL
* No idiopathic urinary calcium stone disease

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* No prior hormonal therapy for prostate cancer
* No concurrent hormonal therapy, including luteinizing hormone-releasing hormone agonists, antiandrogens, glucocorticoids, ketoconazole, finasteride, diethylstilbestrol, or progestins

Radiotherapy:

* No prior brachytherapy or external beam radiotherapy for prostate cancer

Surgery:

* See Disease Characteristics

Other:

* At least 7 days since prior vitamin D therapy or calcium supplements
* No other concurrent vitamin D analogues or calcium supplements
* No concurrent magnesium-containing antacids
* No concurrent thiazide-containing diuretics
* No concurrent phenytoin, phenobarbital, glutethimide, digoxin, or digitalis

Ages: 21 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2001-08; Primary Completion 2006-02 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Intermediate endpoint biomarker modulation | 18 months
Toxicity | 30 months

CONTACTS AND LOCATIONS:
Overall Officials: George Wilding, MD, Study Chair — University of Wisconsin, Madison
Locations (6):
- United States (6):
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Veterans Affairs Medical Center - Madison, Madison, Wisconsin
  - Meriter Hospital, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/